CLINICAL TRIAL: NCT03687892
Title: Establishing Functional Biomarkers for Spaced Theta-Burst Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study personnel.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Instructor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 39234
Record Dates: First submitted 2016-11-08; First posted 2018-09-27 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: repetitive Transcranial Magnetic Stimulation; functional MRI; Theta Burst Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- continuous Theta Burst Stimulation (Experimental): The investigators will perform two applications of 40s of continuous Theta Burst Stimulation (cTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left motor cortex will be determined by Localite Neuronavigation. The baseline structural scan obtained during the scan 1 will be utilized for this localization process.
  Interventions: Device: continuous Theta Burst Stimulation
- intermittent Theta Burst Stimulation (Experimental): The investigators will perform two applications of 40s of intermittent Theta Burst Stimulation (iTBS) form of rTMS at 80% resting motor threshold (previously determined), with a 15 minute intersession interval. The standardized treatment location for the left motor cortex will be determined by Localite Neuronavigation. The baseline structural scan obtained during the scan 1 will be utilized for this localization process.
  Interventions: Device: intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: continuous Theta Burst Stimulation — Continuous Theta Burst Simulation will be applied in a continuous manner resulting in cortical excitability.
  Other Names: cTBS
  Arms: continuous Theta Burst Stimulation
Device: intermittent Theta Burst Stimulation — Intermittent Theta Burst Stimulation will be applied in an intermittent manner resulting in cortical inhibition.
  Other Names: iTBS
  Arms: intermittent Theta Burst Stimulation

SUMMARY:
The investigators plan to use functional magnetic resonance imaging (fMRI) methods to assess brain changes following spaced theta burst stimulation (TBS), a new form of repetitive transcranial magnetic stimulation (rTMS), in 10 healthy participants. The investigators will measure the effects of both excitatory (intermittent, iTBS) and inhibitory (continuous, cTBS) TBS applied to the motor cortex, a system that when stimulated produces a readily observable behavioral response (e.g., movement of a given body regions). In addition to brain activity, we will assess the effects of TBS on motor responses and pain perception. The goal is to determine how brain activity and blood flow during tasks and at rest change following the applications of spaced cTBS and iTBS. Additionally, the aim is to determine the duration of the spaced TBS effects on brain activity and behavior. This study will provide an understanding of the functional brain and behavioral changes that occur following spaced TBS to the motor cortex and has implications for reducing the long treatment schedules associated with classical rTMS protocols.

DETAILED DESCRIPTION:
Overall study design:

The investigators propose a functional MRI study of 10 healthy participants recruited from the community using a cross-over design over two days. On day 1, half of the participants will be randomized to receive iTBS and half will receive cTBS. On scan day 2 the alternate form of TBS will be applied such that all participants will have completed iTBS and cTBS sessions at the end of the two study days.

MRI scan days 1 and 2 will be identical except that iTBS will be applied on one day and cTBS on the other. The duration of the MRI scan session will be approximately 120 minutes each day. The iTBS and cTBS scans sessions will be separated by at least 3 days to ensure that the effects of scan day 1 are not carried over to scan day 2.

Each scan day will consist of the following sessions:

1. Pre-scan session
2. Baseline scan
3. TBS (individually targeted to M1)
4. Post-TBS scan

Participants and Screening:

10 healthy individuals from the community will be recruited. Potential participants will be screened using the MRI Safety Screening Questionnaire, the Transcranial Magnetic Stimulation Adult Safety Screen (TASS), and the Mini Mental State Examination (MMSE) to exclude individuals with contraindications to MRI, TMS, or with cognitive impairments, respectively. Eligible participants will provide written informed consent.

Experimental Design:

Participants will be asked to refrain from taking any analgesic medication for 24 hours prior to scan days. At the start of each scan day, participants will first undergo a Pre-scan session outside of the scanner. In this session, baseline resting motor thresholds and pain thresholds to laser stimuli will be obtained. Participants will also have the opportunity to practice the motor and pain tasks that they will perform in the MRI sessions during this time. For the motor task participants will be asked to tap their finger when a verbal and/or auditory cue is provided. For the pain task, participants will passively experience and rate laser stimuli applied to different regions of the dorsum of their fingers/hands using a 0-10 numerical rating scale (NRS). Ratings will be made for both pain intensity and pain unpleasantness.

On both scan days (iTBS and cTBS) baseline MRI scans will be acquired. These scans will include the following: a high-resolution anatomical scan, a resting-state scan, a motor task scan, a pain task scan, cerebral blood flow imaging, and an interleaved TMS-fMRI scan.

Participants will then be removed from the scanner and receive a spaced TBS session (either iTBS or cTBS depending on the day) whereby 2 TBS protocols are applied with a 15 minute break in between. TBS will be applied at The stimulation will be delivered at 90% of the resting motor threshold. The brain region that will be targeted is the M1 region with the highest activity from the fMRI motor task that occurred in the baseline scan. In this way, each participant will receive TBS that is individually targeted based on their brain function.

Following TBS, participants will then receive their post-TBS MRI scans as described in the baseline scan session.

Study Specifics:

rTMS administration: Using single pulse TMS the scalp position of lowest motor threshold for the right first dorsal interosseous or abductor pollicis brevis muscles will be determined. Resting motor threshold (rMT) will be defined by the lowest power setting producing a visible muscle contraction in 50% trials utilizing PEST software. The investigators will then perform 40 seconds of cTBS or iTBS (depending on the session), which will be followed by 15 minutes of spacing, and then an additional 40 seconds of cTBS or iTBS as has been previously described. The individualized TBS target location for the left M1 will be determined by using each participants' functional motor task MRI scan and Localite Neuronavigation. The baseline structural scan obtained during scan 1 will also be utilized for this localization process.

Pain induction assessment procedures: On the scanning days, baseline warmth sensation threshold, heat-pain threshold (HPTpre) and suprathreshold stimulus intensities and maximum heat tolerance temperature (HTTpre) will be determined for each volunteer using an MRI-safe infrared diode laser stimulator. A 1.5 s, heating ramp up to 20 °C/s will be applied to 10-20 spots (40 mm2) on the hairy skin of the hand and fingers (but not the thumb) of participants.

Pain threshold will be determined using a random staircase method of assessment. The average laser power necessary to produce a rating of "1" will be used to establish the pain threshold. To determine an intensity-effect relationship, pulses will then applied with increasing stimulus intensities to different areas of the dorsum of the hand/fingers with at least 30 s between stimuli. Subjects will be asked to rate the pain intensity and unpleasantness immediately after each stimulus (0 to 10, NRS).

Stimulus intensities will be increased in 300 mW increments. Intensity increases will be continued until a given subject reports a level of moderate pain intensity (5 out of 10, NRS). This intensity will be considered "suprathreshold" for the scan studies. In order to train volunteers in rating their pain with an 11-point numerical rating scale (0 to 10, NRS), the temperature of the laser will then be set to evoke random skin temperatures for 5 s between the individual HPTpre and HTTpre separated by 30-s intervals, and the volunteers were asked to rate their pain. For scans after rTMS-augmented hypnotic analgesia or hypnotic analgesia alone (sham rTMS + hypnotic analgesia), heat pain scores evoked by the pre-established threshold and suprathreshold laser powers will be assessed following each scan. Decreased pain ratings will determine the strength of any analgesic effect TBS. Subjects will be asked to rate their laser-evoked pain following each stimulus during each scan.

Physiologic data acquisition: Throughout the scanning procedure we will monitor peripheral autonomic physiology using MRI compatible EKG leads and a chest belt that monitors respiration. This will allow us to compute respiratory sinus arrhythmia, which provides a good estimate of vagal tone, which, in turn, is associated with better cardiac health and self-soothing. Customized algorithms developed here at Stanford for simultaneous fMRI/EEG to remove MRI scanner artifact from the EKG tracing will be applied.

Brain Imaging Scans:

1. T1-weighted scan (high-resolution anatomical image)
2. Resting-state scan
3. BOLD motor-tapping task scan
4. Pain task scan
5. Arterial-spin labeling scan (cerebral blood flow)
6. Interleaved TMS-fMRI scan

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Right-handed
* Agree to having fMRI scan
* Willingness to suspend use of analgesic drugs or cough suppressants for 24 hours prior to the scans
* Proficiency in English sufficient to complete questionnaires/follow instructions during fMRI assessments
* US Citizen or resident able to receive payment legally

Exclusion Criteria:

* A medical condition that would contraindicate the use of rTMS
* Any condition that would contraindicate MRI (like ferromagnetic metal in the body)
* Pregnancy or breast feeding
* Any significant neurologic disease, including dementia, multi-infarct dementia, Parkinson's or Huntington's disease, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of significant head trauma
* Current antidepressant use (must be washed out for two weeks prior to starting protocol)
* Inability to stop taking medication contraindicated with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Background] Barker AT, Jalinous R, Freeston IL. Non-invasive magnetic stimulation of human motor cortex. Lancet. 1985 May 11;1(8437):1106-7. doi: 10.1016/s0140-6736(85)92413-4. No abstract available. PMID 2860322
- [Background] Alexander GE, DeLong MR, Strick PL. Parallel organization of functionally segregated circuits linking basal ganglia and cortex. Annu Rev Neurosci. 1986;9:357-81. doi: 10.1146/annurev.ne.09.030186.002041. No abstract available. PMID 3085570
- [Background] George MS, Taylor JJ, Short EB. The expanding evidence base for rTMS treatment of depression. Curr Opin Psychiatry. 2013 Jan;26(1):13-8. doi: 10.1097/YCO.0b013e32835ab46d. PMID 23154644
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Baeken C, Marinazzo D, Wu GR, Van Schuerbeek P, De Mey J, Marchetti I, Vanderhasselt MA, Remue J, Luypaert R, De Raedt R. Accelerated HF-rTMS in treatment-resistant unipolar depression: Insights from subgenual anterior cingulate functional connectivity. World J Biol Psychiatry. 2014 May;15(4):286-97. doi: 10.3109/15622975.2013.872295. Epub 2014 Jan 21. PMID 24447053
- [Background] Baeken C, Marinazzo D, Everaert H, Wu GR, Van Hove C, Audenaert K, Goethals I, De Vos F, Peremans K, De Raedt R. The Impact of Accelerated HF-rTMS on the Subgenual Anterior Cingulate Cortex in Refractory Unipolar Major Depression: Insights From 18FDG PET Brain Imaging. Brain Stimul. 2015 Jul-Aug;8(4):808-15. doi: 10.1016/j.brs.2015.01.415. Epub 2015 Feb 7. PMID 25744500
- [Background] Liston C, Chen AC, Zebley BD, Drysdale AT, Gordon R, Leuchter B, Voss HU, Casey BJ, Etkin A, Dubin MJ. Default mode network mechanisms of transcranial magnetic stimulation in depression. Biol Psychiatry. 2014 Oct 1;76(7):517-26. doi: 10.1016/j.biopsych.2014.01.023. Epub 2014 Feb 5. PMID 24629537
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Larson J, Lynch G. Induction of synaptic potentiation in hippocampus by patterned stimulation involves two events. Science. 1986 May 23;232(4753):985-8. doi: 10.1126/science.3704635.
- [Background] Suppa A, Huang YZ, Funke K, Ridding MC, Cheeran B, Di Lazzaro V, Ziemann U, Rothwell JC. Ten Years of Theta Burst Stimulation in Humans: Established Knowledge, Unknowns and Prospects. Brain Stimul. 2016 May-Jun;9(3):323-335. doi: 10.1016/j.brs.2016.01.006. Epub 2016 Jan 27. PMID 26947241
- [Background] Cao G, Harris KM. Augmenting saturated LTP by broadly spaced episodes of theta-burst stimulation in hippocampal area CA1 of adult rats and mice. J Neurophysiol. 2014 Oct 15;112(8):1916-24. doi: 10.1152/jn.00297.2014. Epub 2014 Jul 23. PMID 25057146
- [Background] Goldsworthy MR, Pitcher JB, Ridding MC. Spaced Noninvasive Brain Stimulation: Prospects for Inducing Long-Lasting Human Cortical Plasticity. Neurorehabil Neural Repair. 2015 Sep;29(8):714-21. doi: 10.1177/1545968314562649. Epub 2014 Dec 11. PMID 25505220
- [Background] Nyffeler T, Cazzoli D, Hess CW, Muri RM. One session of repeated parietal theta burst stimulation trains induces long-lasting improvement of visual neglect. Stroke. 2009 Aug;40(8):2791-6. doi: 10.1161/STROKEAHA.109.552323. Epub 2009 Jun 11. PMID 19520986
- [Background] Cazzoli D, Muri RM, Schumacher R, von Arx S, Chaves S, Gutbrod K, Bohlhalter S, Bauer D, Vanbellingen T, Bertschi M, Kipfer S, Rosenthal CR, Kennard C, Bassetti CL, Nyffeler T. Theta burst stimulation reduces disability during the activities of daily living in spatial neglect. Brain. 2012 Nov;135(Pt 11):3426-39. doi: 10.1093/brain/aws182. Epub 2012 Jul 24. PMID 22831781
- [Background] Nyffeler T, Wurtz P, Luscher HR, Hess CW, Senn W, Pflugshaupt T, von Wartburg R, Luthi M, Muri RM. Extending lifetime of plastic changes in the human brain. Eur J Neurosci. 2006 Nov;24(10):2961-6. doi: 10.1111/j.1460-9568.2006.05154.x. PMID 17156218
- [Background] Goldsworthy MR, Pitcher JB, Ridding MC. Neuroplastic modulation of inhibitory motor cortical networks by spaced theta burst stimulation protocols. Brain Stimul. 2013 May;6(3):340-5. doi: 10.1016/j.brs.2012.06.005. Epub 2012 Jul 5. PMID 22835528
- [Background] Goldsworthy MR, Pitcher JB, Ridding MC. The application of spaced theta burst protocols induces long-lasting neuroplastic changes in the human motor cortex. Eur J Neurosci. 2012 Jan;35(1):125-34. doi: 10.1111/j.1460-9568.2011.07924.x. Epub 2011 Nov 25. PMID 22118241
- [Background] Duprat R, Desmyter S, Rudi de R, van Heeringen K, Van den Abbeele D, Tandt H, Bakic J, Pourtois G, Dedoncker J, Vervaet M, Van Autreve S, Lemmens GM, Baeken C. Accelerated intermittent theta burst stimulation treatment in medication-resistant major depression: A fast road to remission? J Affect Disord. 2016 Aug;200:6-14. doi: 10.1016/j.jad.2016.04.015. Epub 2016 Apr 19. PMID 27107779
- [Background] Koch G, Bonni S, Giacobbe V, Bucchi G, Basile B, Lupo F, Versace V, Bozzali M, Caltagirone C. theta-burst stimulation of the left hemisphere accelerates recovery of hemispatial neglect. Neurology. 2012 Jan 3;78(1):24-30. doi: 10.1212/WNL.0b013e31823ed08f. Epub 2011 Dec 14. PMID 22170878
- [Background] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188
- [Background] Larson J, Munkacsy E. Theta-burst LTP. Brain Res. 2015 Sep 24;1621:38-50. doi: 10.1016/j.brainres.2014.10.034. Epub 2014 Oct 27. PMID 25452022
- [Background] Siebner HR, Takano B, Peinemann A, Schwaiger M, Conrad B, Drzezga A. Continuous transcranial magnetic stimulation during positron emission tomography: a suitable tool for imaging regional excitability of the human cortex. Neuroimage. 2001 Oct;14(4):883-90. doi: 10.1006/nimg.2001.0889. PMID 11554807
- [Background] Fox P, Ingham R, George MS, Mayberg H, Ingham J, Roby J, Martin C, Jerabek P. Imaging human intra-cerebral connectivity by PET during TMS. Neuroreport. 1997 Aug 18;8(12):2787-91. doi: 10.1097/00001756-199708180-00027. PMID 9295118
- [Background] Siebner HR, Peller M, Willoch F, Minoshima S, Boecker H, Auer C, Drzezga A, Conrad B, Bartenstein P. Lasting cortical activation after repetitive TMS of the motor cortex: a glucose metabolic study. Neurology. 2000 Feb 22;54(4):956-63. doi: 10.1212/wnl.54.4.956. PMID 10690992
- [Background] Bohning DE, Shastri A, Nahas Z, Lorberbaum JP, Andersen SW, Dannels WR, Haxthausen EU, Vincent DJ, George MS. Echoplanar BOLD fMRI of brain activation induced by concurrent transcranial magnetic stimulation. Invest Radiol. 1998 Jun;33(6):336-40. doi: 10.1097/00004424-199806000-00004. PMID 9647445
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Subthreshold high-frequency TMS of human primary motor cortex modulates interconnected frontal motor areas as detected by interleaved fMRI-TMS. Neuroimage. 2003 Nov;20(3):1685-96. doi: 10.1016/j.neuroimage.2003.07.028. PMID 14642478
- [Background] Bohning DE, Shastri A, McConnell KA, Nahas Z, Lorberbaum JP, Roberts DR, Teneback C, Vincent DJ, George MS. A combined TMS/fMRI study of intensity-dependent TMS over motor cortex. Biol Psychiatry. 1999 Feb 15;45(4):385-94. doi: 10.1016/s0006-3223(98)00368-0. PMID 10071706
- [Background] Speer AM, Willis MW, Herscovitch P, Daube-Witherspoon M, Shelton JR, Benson BE, Post RM, Wassermann EM. Intensity-dependent regional cerebral blood flow during 1-Hz repetitive transcranial magnetic stimulation (rTMS) in healthy volunteers studied with H215O positron emission tomography: II. Effects of prefrontal cortex rTMS. Biol Psychiatry. 2003 Oct 15;54(8):826-32. doi: 10.1016/s0006-3223(03)00324-x. PMID 14550682
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Functional MRI of the immediate impact of transcranial magnetic stimulation on cortical and subcortical motor circuits. Eur J Neurosci. 2004 Apr;19(7):1950-62. doi: 10.1111/j.1460-9568.2004.03277.x. PMID 15078569
- [Background] Chouinard PA, Van Der Werf YD, Leonard G, Paus T. Modulating neural networks with transcranial magnetic stimulation applied over the dorsal premotor and primary motor cortices. J Neurophysiol. 2003 Aug;90(2):1071-83. doi: 10.1152/jn.01105.2002. Epub 2003 Apr 17. PMID 12702714
- [Background] Nettekoven C, Volz LJ, Kutscha M, Pool EM, Rehme AK, Eickhoff SB, Fink GR, Grefkes C. Dose-dependent effects of theta burst rTMS on cortical excitability and resting-state connectivity of the human motor system. J Neurosci. 2014 May 14;34(20):6849-59. doi: 10.1523/JNEUROSCI.4993-13.2014. PMID 24828639
- [Background] Cardenas-Morales L, Gron G, Kammer T. Exploring the after-effects of theta burst magnetic stimulation on the human motor cortex: a functional imaging study. Hum Brain Mapp. 2011 Nov;32(11):1948-60. doi: 10.1002/hbm.21160. Epub 2010 Dec 22. PMID 21181786
- [Background] Orosz A, Jann K, Wirth M, Wiest R, Dierks T, Federspiel A. Theta burst TMS increases cerebral blood flow in the primary motor cortex during motor performance as assessed by arterial spin labeling (ASL). Neuroimage. 2012 Jul 2;61(3):599-605. doi: 10.1016/j.neuroimage.2012.03.084. Epub 2012 Apr 12. PMID 22613775
- [Background] Watanabe T, Hanajima R, Shirota Y, Ohminami S, Tsutsumi R, Terao Y, Ugawa Y, Hirose S, Miyashita Y, Konishi S, Kunimatsu A, Ohtomo K. Bidirectional effects on interhemispheric resting-state functional connectivity induced by excitatory and inhibitory repetitive transcranial magnetic stimulation. Hum Brain Mapp. 2014 May;35(5):1896-905. doi: 10.1002/hbm.22300. Epub 2013 Jul 29. PMID 23897535
- [Background] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Continuous or intermittent Theta Burst Stimulation (iTBS). No participants were randomized to treatment so data are presented in one group.
Period: Overall Study
Arm/Group | All Participants
Started | 37
Completed | 0
Not Completed | 37

BASELINE CHARACTERISTICS:
Population: Participants who were consented and received baseline scan.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.77 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Changes in Motor Evoked Potential
Description: To determine the duration of effect of an application of a spaced TBS stimulation session (both inhibitory, cTBS and excitatory, iTBS) as measured by duration of change in motor evoked potential.
Time Frame: Prior to and and immediately after TBS sessions on each day (separated by 3+ days)
Population: No outcome measure analysis was possible because no post-baseline data were collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline Resting-state Functional Connectivity Between the M1 Hotspot and Other Motor Areas Immediately Post-TBS
Description: To determine the resting state functional connectivity changes that result from an application of spaced TBS stimulations (both inhibitory, cTBS and excitatory, iTBS).
Time Frame: Prior to and and immediately after TBS sessions on each day (separated by 3+ days)
Population: No outcome measure analysis was possible because no post-baseline data were collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline Motor Cortex Activity as Assessed by the BOLD Signal Immediately Post-TBS
Description: To determine the TMS-BOLD (over M1) changes that result from an application of spaced TBS stimulations (both inhibitory, cTBS and excitatory, iTBS).
Time Frame: Prior to and and immediately after TBS sessions on each day (separated by 3+ days)
Population: No outcome measure analysis was possible because no post-baseline data were collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Arterial Perfusion
Description: To determine the arterial perfusion changes that result from an application of spaced TBS stimulations (both inhibitory, cTBS and excitatory, iTBS) as measured by ASL.
Time Frame: Prior to and and immediately after TBS sessions on each day (separated by 3+ days)
Population: No outcome measure analysis was possible because no post-baseline data were collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-10-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT03687892/Prot_000.pdf